CLINICAL TRIAL: NCT07356037
Title: A Prospective Clinical Study of Nanocrystalline Megestrol Acetate in Combination With Standard Therapy Versus Standard Therapy Alone for Cachectic Stage Locally Advanced Hepatocellular Carcinoma
Brief Title: Nanocrystalline Megestrol Acetate for Cachectic Stage Locally Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EpiCure-HCC 01
Record Dates: First submitted 2026-01-04; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cachexia; Hepatocellular Carcinoma
MeSH Terms: conditions — Cachexia; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanocrystalline Megestrol Acetate Oral Suspension + Standard Antitumor Therapy (Experimental): Nanocrystalline Megestrol Acetate Oral Suspension + Standard Antitumor Therapy
  Interventions: Drug: Nanocrystalline Megestrol Acetate; Combination Product: Standard Antitumor Therapy
- Standard Antitumor Therapy (Active Comparator): Standard Antitumor Therapy
  Interventions: Combination Product: Standard Antitumor Therapy

INTERVENTIONS:
Drug: Nanocrystalline Megestrol Acetate — Nanocrystalline Megestrol Acetate oral suspension, with a specification of 125 mg/mL, administered orally at a dose of 5 mL per day (625 mg/day), and the primary endpoint efficacy collection will be conducted in the 4th week.
  Arms: Nanocrystalline Megestrol Acetate Oral Suspension + Standard Antitumor Therapy
Combination Product: Standard Antitumor Therapy — Standard Antitumor Therapy

SUMMARY:
This study is a prospective, randomized, parallel-controlled clinical trial. The primary objective is to evaluate the superiority and safety of nanocrystalline megestrol acetate in combination with standard therapy compared with standard therapy alone in improving appetite and body mass index (BMI) during treatment in patients with early-stage or locally advanced hepatocellular carcinoma at the cachexia stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hepatocellular carcinoma who have not previously received systemic therapy and are confirmed by histological or cytological assessment, as evaluated by the investigator, to be unsuitable or ineligible for curative surgical resection; Barcelona Clinic Liver Cancer (BCLC) stage B-C.
2. Child-Pugh class A or B7.
3. Planned to receive interventional therapy in combination with systemic antitumor therapy.
4. At least one measurable tumor lesion according to mRECIST v1.1.
5. Meet the diagnostic criteria for pre-cachexia or cachexia (based on the Fearon criteria).

Exclusion Criteria:

1. Presence of any condition affecting gastrointestinal absorption, such as dysphagia, malabsorption, or uncontrolled vomiting; patients receiving tube feeding or parenteral nutrition.
2. Presence of anorexia due to anorexia nervosa, psychiatric disorders, or pain that makes eating difficult.
3. Patients with acquired immunodeficiency syndrome (AIDS).
4. Currently receiving or planning to receive other medications that increase appetite or body weight, such as corticosteroids (except short-term dexamethasone during chemotherapy), androgens, progestins, thalidomide, olanzapine, anamorelin, or other appetite stimulants.
5. Patients with Cushing's syndrome, adrenal or pituitary insufficiency, or poorly controlled diabetes mellitus.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with improved appetite based on A/CS-12 assessment. | The proportion of subjects with improved appetite based on A/CS-12 assessment in 12 weeks

SECONDARY OUTCOMES:
Proportion of patients with BMI increase | Proportion of patients with BMI increase in 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan, China